CLINICAL TRIAL: NCT07074587
Title: Investigation of the Effects of Spinal Stabilization Exercises Focusing on the Pelvic Floor on Core Stability, Urinary Symptoms, and Pelvic Floor Muscle Function in Women With Multiple Sclerosis and Lower Urinary Tract Symptoms
Brief Title: Effects of Spinal Stabilization on the Pelvic Floor in Women With Multiple Sclerosis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Gözde TEKİN, Phd, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AİBU-FTR-GT-001
Record Dates: First submitted 2025-06-25; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis; Urinary Incontinence; Lower Urinary Tract Symptoms
Keywords: Multiple Sclerosis; Lower Urinary Tract Symptoms; Urinary Incontinence; Core Stability; Spinal Stabilization
MeSH Terms: conditions — Multiple Sclerosis; Urinary Incontinence; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to a control group that receives pelvic floor muscle exercises only or an experimental group that receives both pelvic floor muscle exercises and spinal stabilization exercise focused on the pelvic floor.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to group allocation to minimize bias during post-intervention evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic floor muscle exercises (Active Comparator): Pelvic floor muscle exercises will be taught with an innovative approach based on the principles of finding, feeling, forcing, following and functional training of the pelvic floor muscles. Pelvic floor muscle exercises will be applied as 3 sets in the first 2 weeks, 4 sets in the 3rd and 4th weeks, 5 sets in the 5th and 6th weeks, and finally 6 sets in the 7th and 8th weeks. Individuals will continue their pelvic floor muscle exercises as a home program.
  Interventions: Behavioral: Pelvic floor muscle exercises
- Spinal stabilization exercises focusing on the pelvic floor + Pelvic floor muscle exercises (Experimental): Spinal stabilization exercises focusing on the pelvic floor will be administered under physiotherapist supervision three times per week for eight weeks. Each session will consist of 5 minutes of warm-up, 30 minutes of pelvic floor-focused spinal stabilization exercises, and 5 minutes of cool-down. Stabilization and posture training will be provided at the outset, including instruction on identifying the neutral position of the spine to ensure proper posture. Correct pelvic floor muscle contraction and abdominal bracing techniques will be demonstrated. The exercise program will comprise three phases: static (weeks 1-2), dynamic (weeks 3-5), and functional (weeks 6-8). Throughout all exercises, participants will maintain a neutral spine position and abdominal bracing, with contractions held for 5-10 seconds and repeated 10 times. Additionally, participants will be instructed to continue pelvic floor exercises as a home program on non-supervised days.
  Interventions: Behavioral: Spinal stabilization exercises focusing on the pelvic floor + Pelvic floor muscle exercises

INTERVENTIONS:
Behavioral: Pelvic floor muscle exercises — Pelvic floor muscle exercises will be taught with an innovative approach based on the principles of finding, feeling, forcing, following and functional training of the pelvic floor muscles. Pelvic floor muscle exercises will be applied as 3 sets in the first 2 weeks, 4 sets in the 3rd and 4th weeks, 5 sets in the 5th and 6th weeks, and finally 6 sets in the 7th and 8th weeks. Individuals will continue their pelvic floor muscle exercises as a home program.
  Arms: Pelvic floor muscle exercises
Behavioral: Spinal stabilization exercises focusing on the pelvic floor + Pelvic floor muscle exercises — This program consists of 3 phases: 30 minutes of spinal stabilization exercises focusing on the pelvic floor, 5 minutes of warm-up and 5 minutes of cool-down exercises.The exercises will consist of 3 phases: static, dynamic and functional phases. Individuals will perform static phase exercises for the first 2 weeks, then dynamic phase exercises in the 3rd and 5th weeks and finally functional phase exercise in the 6th and 8th weeks. Individuals will be asked to maintain neutral spine position and abdominal bracing during pelvic floor muscle contraction during all exercises. Individuals will maintain the contraction for 5-10 seconds for 10 repetitions in each position in all phases.
  Arms: Spinal stabilization exercises focusing on the pelvic floor + Pelvic floor muscle exercises

SUMMARY:
The purpose of this study was to investigate the effects of spinal stabilization exercises focusing on the pelvic floor on core stability, urinary symptoms and pelvic floor muscle function in women with Multiple Sclerosis and lower urinary tract symptoms. Participants will be randomly assigned to a control group that receives pelvic floor muscle exercises only or an experimental group that receives both pelvic floor muscle exercises and spinal stabilization exercise focused on the pelvic floor. Outcome measures will be assessed pre- and post-intervention using validated instruments.

DETAILED DESCRIPTION:
In multiple sclerosis (MS), disruption of the neural pathways responsible for bladder control leads to the development of lower urinary tract symptoms (LUTS). These symptoms, observed in approximately 32-96% of individuals with MS, have a significant negative impact on quality of life. Conservative management of LUTS includes lifestyle modifications, bladder training, and pelvic floor muscle training (PFMT). Although the effectiveness of PFMT has been demonstrated, there is no standardized protocol regarding exercise type or duration, indicating a gap in the literature concerning the identification of the most effective approach. Moreover, existing studies emphasize that the effective contraction of pelvic floor muscles requires the simultaneous activation of deep core muscles, particularly the transversus abdominis. This suggests that pelvic floor rehabilitation without the involvement of abdominal muscles may be insufficient. Spinal stabilization exercises target deep core muscles to enhance neuromuscular control, strength, and endurance. Recently, "spinal stabilization exercises focusing on the pelvic floor" have emerged as a promising strategy in the management of urinary incontinence. However, research on trunk control in individuals with MS remains limited and primarily focuses on neurological symptoms, with minimal attention given to LUTS and pelvic floor function.

This study is designed as a prospective, randomized controlled trial to evaluate the effects of spinal stabilization exercises focusing on the pelvic floor, delivered in addition to PFMT, on core stability, urinary symptoms, and pelvic floor muscle function in women with MS and LUTS. Eligible participants who consent to join the study will be randomly allocated into two groups using block randomization. The control group will receive PFMT alone, while the experimental group will receive PFMT combined with spinal stabilization exercises focusing on the pelvic floor . Both interventions will be delivered three times per week for eight weeks. Primary and secondary outcomes will be assessed using validated objective and subjective tools at baseline and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged between 18 and 65 years
* Being diagnosed with Multiple Sclerosis by a specialist neurologist and having lower urinary system symptoms [Overactive Bladder-V8 scale score ≥ 9 and having at least two of the lower urinary system symptoms (urinary incontinence, nocturia, daytime urination frequency >8, storage symptoms such as sudden feeling of tightness, intermittent urination, slow urine flow and emptying symptoms such as incomplete emptying)
* Being in the mild or moderate stage of the disease (Expanded Disability Status Scale (EDSS) score ˂ 6
* No relapse experienced within the past month
* Scoring 24 or above on the Mini-Mental State Examination (MMSE)
* Being literate
* Willingness to voluntarily participate in the study
* Ability to perform voluntary pelvic floor muscle contractions
* No changes in medical treatment within the past three months
* Ability to understand and cooperate with the assessments and interventions involved in the study

Exclusion Criteria:

* Diagnosis of one or more neurological disorders other than Multiple Sclerosis
* Body mass index (BMI) ≥ 30
* Diagnosis of overflow urinary incontinence
* History of antimuscarinic medication use
* Presence of advanced pelvic organ prolapse (stage ≥ 2)
* Active urinary tract infection
* History of cesarean section or vaginal delivery within the past 6 months
* Diagnosis of any other neurological condition that may cause urinary incontinence
* History of urological or gynecological surgery
* History of malignancy
* Currently pregnant or not sexually active (coitus negative)
* Participation in exercise training or physical therapy for lower urinary tract symptoms within the past 6 months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Urinary Symptoms | 8 week
  Urinary symptoms will be assessed with the International Incontinence Questionnaire Short Form. The International Incontinence Questionnaire Short Form consists of a total of six questions. The total score is obtained by summing the scores of questions 3, 4 and 5. Scores that can be obtained from the scale vary between 0-21; a low score indicates that urinary incontinence affects quality of life a little, while a high score indicates that it affects it a lot.
Evaluation of Bladder Functions | 8 week
  A bladder diary will be used to assess bladder function for lower urinary tract symptoms. Patients will be asked to complete a 24-hour bladder diary on three non-consecutive days. Average day-night voiding frequency, voiding volume and number of urinary incontinence will be calculated by averaging the three daily urinary diaries.

SECONDARY OUTCOMES:
Evaluation of the degree of urinary symptoms | 8 week
  Overactive Bladder-Version8 will be used to assess the degree of lower urinary system symptoms due to overactive bladder. The score to be obtained from the scale ranges from "0" the best to "40" the worst. If the total score on the scale is more than 8, the subjects are considered to have possible lower urinary tract symptoms.
Evaluation of Pelvic Floor Muscle Function | 8 week
  Pelvic floor muscle function will be evaluated with the 632 Myomed biofeedback device. The pressure probe and device will be disinfected in each individual before the application and the probe will be used with a condom to ensure the hygiene of the individual. During the assessment, the pressure probe will be inserted intravaginally while the individual is supine, knees bent and slightly apart. Assessment results will be recorded in hectopascal.
Evaluation of pelvic floor muscle strength | 8 week
  Vaginal palpation method will be used to measure pelvic floor muscle strength. The assessment will be performed in supine position, with hips and knees flexed and soles of the feet in contact with the bed. After taking the necessary hygiene measures, the physiotherapist will place the index and middle finger intravaginally. The individual will then be asked to pinch the physiotherapist's fingers and pull upwards for pelvic floor muscle contraction. The outcome value will be scored with the Modified Oxford grading system.
Evaluation of the endurance of the lateral core muscles | 8 week
  The lateral bridge test will be used to assess the endurance of the lateral core muscles. Individuals will be asked to place their forearms and feet on the side of one side in a position to carry their body weight, then they will be asked to maintain this position by lifting their hips from the bed. The test will be terminated when the proper posture is broken or the pelvis falls on the bed, and the time from maintaining the proper position to breaking the position will be recorded in seconds. The test will be performed separately on the right and left side.
Evaluation of the endurance of the anterior core muscles | 8 week
  Flexor endurance test will be used to assess the endurance of the anterior core muscles. Individuals will be placed on the bed with their trunk at 60°, knees and hips at 90° flexion and supported by their feet. In this position, the time in seconds will be recorded until they lose 60° of trunk flexion.
Evaluation of endurance of the posterior core muscles | 8 week
  The extensor endurance test will be used to evaluate the endurance of the posterior core muscles. Individuals will lie in a prone position with pelvis, hips and knees supported on the bed and the upper trunk will be positioned on the edge of the bed in a straight, slightly extended position. Individuals will be stabilized by their feet. The test will be terminated when the trunk falls from the horizontal position to flexion and the time in this position will be recorded in seconds.
Evaluation of Deep Lumbar Muscular Strength | 8 week
  Stabilizer Pressure Biofeedback device will be used to assess deep lumbar muscular strength. Individuals will be asked to lie in a prone position and keep their knees in a straight position, their spine straight and their head in a comfortable position. The cushion of the measuring device will be placed under their abdominal area with the air completely deflated. After the manometer needle is set to 70 mm/Hg, the individuals will be asked to contract the transversus abdominous muscles for 5 seconds as taught. The test will be performed for 10 s and 3 repetitions and the average of the results of the 3 tests will be recorded in mm/Hg.
Evaluation of Quality of Life | 8 week
  King Health Questionnaire will be used to assess quality of life. The questionnaire consists of two parts and includes 32 items. . On the complaint severity scale, the best score is "0" and the worst score is "30". In other subsections of the King Health Questionnaire, the best score is "0" and the worst score is "100".
Evaluation of Subjective Perception of Recovery | 8 week
  The Global Perceived Impact scale will be used to assess the subjective perception of improvement after the training. Participants will be asked to rate on a scale of 1 to 9 the extent to which their complaints have improved compared to before the training. The description of the scores is; '1' 'much improved', '2' 'much improved', '3' 'moderately improved', '4' 'slightly improved', '5' 'unchanged', '6' 'slightly worsened', '7' 'moderately worsened', '8' 'much worsened', '9' 'much worsened'.
Evaluation of Perceived Health Problem | 8 week
  The health problem perceived by individuals will be assessed with the Patient-specific complaints instrument. The numbered classification scale-11 (0-10) will be used for scoring. The individual will be asked to give a score between 0-10 for the severity of the problem caused by lower urinary tract symptoms as perceived by the individual. 0 means "no complaint at all" and 10 means "very severe complaint".
Evaluation of Compliance with Training | 8 week
  The compliance of the individuals with the training will be evaluated using a 10-centimeter visual analog scale. At the end of the study, the individuals in the control and experimental groups will be asked to evaluate the training program given to them by marking the place that best expresses themselves on a 10 cm line between 0 (I did not apply the treatment given at all) and 10 (I applied the treatment given completely). The distance between the marked point and the starting point will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: gözde tekin, Msc, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant İzzet Baysal University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Merkez, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No